CLINICAL TRIAL: NCT03323710
Title: A Phase II Study of Propranolol Plus Sunitinib in First-line Treatment of Metastatic Renal Cell Carcinoma (ProSun Study)
Brief Title: Study of Propranolol Plus Sunitinib in First-line Treatment of Metastatic Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patient recruitment.
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Paweł Chrom, M.D., Military Institute od Medicine National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-001
Record Dates: First submitted 2017-10-22; First posted 2017-10-27 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic; Renal Cell Carcinoma; Kidney Cancer; Sunitinib; Sutent; Tyrosine Kinase Inhibitor; Angiogenesis Inhibitor; Propranolol; Beta-blocker; First-line
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Kidney Neoplasms | interventions — Propranolol; Sunitinib

STUDY DESIGN:
Intervention Model Description: Two-stage optimal Simon design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol plus Sunitinib (Experimental)
  Interventions: Drug: Propranolol; Drug: Sunitinib

INTERVENTIONS:
Drug: Propranolol — Propranolol will be administered orally at a starting dose of 40 mg (one tablet) two times a day (total daily dose of 80 mg). In case of acceptable safety profile, the dose may be increased to 80 mg (two tablets) two times a day (total daily dose of 160 mg) or farther to 80 mg (two tablets) three times a day (total daily dose of 240 mg).
Drug: Sunitinib — Sunitinib will be administered orally at a starting dose of 50 mg once daily, for 4 consecutive weeks, followed by a 2-week rest period (schedule 4/2) to comprise a complete cycle of 6 weeks.The schedule may be changed to 2 weeks on / 1 week off (schedule 2/1) and a daily dose may be reduced to 37.5 mg or 25 mg to decrease the level of toxic side effects.
  Other Names: Sutent

SUMMARY:
The study aims to assess antineoplastic efficacy, safety, influence on quality of life and disease-related stress of propranolol taken in combination with sunitinib in previously untreated metastatic renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Histological diagnosis of clear-cell renal cell carcinoma (RCC) or mixed-type RCC with more than 60% of clear-cell component.
2. Diagnosis of stage IV RCC (primary metastatic or recurrence after surgical procedure).
3. Prior nephrectomy (complete or partial).
4. Presence of measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1.
5. Karnofsky performance status score of 80-100%.
6. Favourable- or intermediate-risk according to Memorial Sloan Kettering Cancer Center criteria.
7. Adequate organ function, including the following:

   1. hepatic: total bilirubin ≤ 2 times the upper limit of normal (excluding patients with Gilbert syndrome), aspartate aminotransferase and alanine aminotransferase ≤ 5 times the upper limit of normal,
   2. renal: serum creatinine ≤ 2 times the upper limit of normal,
   3. bone marrow: absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100000/mm3, hemoglobin ≥ 9.5 g/dl.
8. Normal thyroid function (natural or with supplementation of thyroid hormones) defined as thyroid-stimulating hormone within limits of normal.
9. Age eighteen years or older on the day of consent.
10. Written informed consent prior to study entry.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Prior systemic pharmacotherapy of RCC.
2. Treatment with propranolol within 6 months of study entry.
3. Metastases in central nervous system (patients who had central nervous system metastases that were surgically resected and/or treated with radiotherapy in the past and now are without neurological symptoms, are allowed on protocol).
4. Female patients who are pregnant or breast feeding or adults of reproductive potential who are not using effective birth control methods.
5. Presence of other malignancies (patients with carcinoma in situ of the cervix or basal cell carcinoma of the skin are allowed on protocol).
6. Presence of any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   1. heart failure of New York Heart Association Class III or IV, significant cardiac arrhythmia or any other clinically significant cardiovascular disease,
   2. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of entering the study,
   3. severely impaired respiration as defined as O2 saturation that is ≤ 90% at rest on room air,
   4. uncontrolled diabetes as defined by fasting serum glucose > 1.5 times the upper limit of normal,
   5. ejection fraction less than 40% (measured at echocardiography),
   6. significant liver disease such as cirrhosis, active hepatitis or chronic persistent hepatitis,
   7. active (acute or chronic) infections requiring antimicrobial intervention.
7. Concomitant treatment with:

   1. chronic, systemic corticosteroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed,
   2. strong CYP3A4 inducers/inhibitors: carbamazepine, phenytoin, rifabutin, rifampin, nafcillin, phenobarbital, St John's wort, itraconazole, ketoconazole, erythromycin, clarithromycin, nefazodone.
8. Known allergy/sensitivity to sunitinib and/or propranolol.
9. Galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
10. Immunization with attenuated live vaccines within 30 days of study entry.
11. Human immunodeficiency virus sero-positivity at the study entry or in the past.
12. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sunitinib and/or propranolol (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
13. Presence of active, bleeding diathesis.
14. Major surgery (defined as requiring general anesthesia) and/or significant traumatic injury (requiring > 28 days to heal) within 28 days of the study entry; presence of side effects due to any surgery or probable requirement of major surgery during the course of the study.
15. Present contraindications to propranolol, that include: bronchial asthma, prolonged fasting, acidosis, hypotension (systolic blood pressure less than 90 mmHg, diastolic blood pressure less than 60 mmHg), severe peripheral arterial circulatory disturbance, cardiogenic shock, bradycardia, Prinzmetal's angina, uncontrolled heart failure, second or third degree heart block, untreated phaeochromocytoma, sick sinus syndrome.
16. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 18 months
  Objective Response Rate (ORR) is defined as the percentage of patients who have achieved partial response (PR) or complete response (CR) according to the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 18 months
  Overall Survival (OS) is defined as the time from treatment initiation to death from any cause.
Progression-free Survival (PFS) | Up to 18 months
  Progression-free Survival (PFS) is defined as the time from treatment initiation to the first date of objectively determined progressive disease (PD) according to the RECIST v1.1 or death from any cause, whichever occurred first.
Disease Control Rate (DCR) | Up to 18 months
  Disease Control Rate (DCR) is defined as the percentage of patients who have achieved partial response (PR), complete response (CR) or stable disease (SD) according to the RECIST v1.1.
Safety profile as assessed by Common Terminology Criteria for Adverse Events v4.03 summarized by type, frequency, and severity. | Up to 18 months
  Safety profile as assessed by Common Terminology Criteria for Adverse Events v4.03 summarized by type, frequency, and severity.
Health-related Quality of Life (QoL) | Up to 18 months
  Change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) v3.
  The EORTC QLQ-C30 includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range from 0 to 100. High score for a functional scale represents a high / healthy level of functioning. High score for the global health status / QoL represents a high QoL. High score for a symptom scale / item represents a high level of symptomatology / problems. Scoring these scales include the following steps:
  1. Estimate the average of the items that contribute to the scale (the raw score).
  2. Use the linear transformation to standardise the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Health-related Quality of Life (QoL) | Up to 18 months
  Change from baseline in the Functional Assessment of Cancer Therapy-Kidney Symptom Index - 15.
Disease-related Stress (DRS) | Up to 18 months
  Change from baseline in the 10-point Perceived Stress Scale (PSS).
  The PSS is a validated psychological tool for assessing the perception of stress. Patient responses to all of the 10 questions present in the PSS questionnaire range from 0 to 4. To obtain a total result:
  1. Reverse scores for questions 4, 5, 7, and 8.
  2. Add up scores for each question to get a total result. Individual total scores range from 0 to 40. Higher scores indicate higher perceived stress.
Tumour tissue and serum biomarkers status | Up to 18 months
  Descriptive statistics of selected biomarkers from analysis of patient samples.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Chrom, M.D., Principal Investigator — Military Institute od Medicine National Research Institute
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03323710/Prot_SAP_000.pdf